CLINICAL TRIAL: NCT06644547
Title: (Cost)effectiveness of the Intervention 'Gezond En Goed Met Elkaar'
Acronym: GGME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Iris Koelmans, Principal Investigator, VU University of Amsterdam
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024.0213
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: The Study is Focused on People with Limited Health Literacy; We Are Not Studying a Disease or Condition
Keywords: health literacy; positive health; intervention; Gezond en goed met elkaar

STUDY DESIGN:
Intervention Model Description: Pragmatic stepped-wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention 'Gezond en goed met elkaar' (Experimental): see description of the intervention 'Gezond en goed met elkaar'
  Interventions: Behavioral: Gezond en goed met elkaar
- Control group (No Intervention): Participants do not receive the intervention yet. They have to wait 3 months before they start with the intervention. They will fill out questionnaires at baseline, 3, 6 and 9 months.
- Control group 2 (No Intervention): Participants do not receive the intervention yet. They have to wait 6 months before they start with the intervention. They will fill out questionnaires at baseline, 3, 6 and 9 months.

INTERVENTIONS:
Behavioral: Gezond en goed met elkaar — The intervention 'Gezond en goed met elkaar' focuses on improving (positive) health literacy and literacy. The six domains of "positive health" are the focus of the intervention meetings. This intervention has been made available for citizens of Almere, Zwolle, Gouda, Nunspeet and Leusden through collaboration with these municipalities. Lifestyle coaches working in these municipalities implement the intervention.
  Arms: Intervention 'Gezond en goed met elkaar'

SUMMARY:
The goal of this intervention study is to learn if the intervention can increase positive health and health literacy in people with limited health literacy. The main questions it aims to answer are:

* Does participating in the intervention 'Gezond en goed met elkaar' increase participant's positive health?
* Does participating in the intervention 'Gezond en goed met elkaar' improve health literacy?

Researchers will compare people who participate in the intervention with people who haven't participated in the intervention yet.

Participants will:

* participate in the intervention (3 months)
* fill out questionnaires every 3 months

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* analfabetism
* insufficient language level of Dutch to be able to participate in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Positive Health | From baseline measurement to 9 months later
  Positive Health questionnaire developed by Institute of Positive Health (iPH) 17 items, answered on a 10-point Likert scale
Vitality | From baseline measurement to 9 months later
  SF-12 Vitality (VT) question 6b

SECONDARY OUTCOMES:
Health Literacy | From baseline measurement to 9 months later
  HLS-EU-Q16 adapted to B1 language level For the psychometric analyses of HLS-EU-Q16, each of the 16 questions were coded according to the following: 'very difficult'=1 point, 'fairly difficult'=2 points, 'fairly easy'=3 points or 'very easy'=4 points, giving a total of 16-64 scores. The HLS-EU-Q16 manual recommends dichotomizing the answers from HLS-EU-Q16 ('very difficult'/'fairly difficult'=0, 'fairly easy'/'very easy'=1; total 0-16 scores)
  1 & 2 -> 0 3 & 4 -> 1
  dividing the total scores into three categories of HL: 0-8 = inadequate 9-12 = problematic 13-16 = adequate
Basic Psychological Needs | From baseline measurement to 9 months later
  BPNSFS-ID: Basic Psychological Needs Satisfaction and Frustration Scale
Well-Being | From baseline measurement to 9 months later
  ASCOT: The Adult Social Care Outcomes Toolkit - dutch translation
Quality of Life (QALYs) | From baseline measurement to 9 months later
  EQ-5D-5L: 5-level EQ-5D version (EuroQol Group, 2009)
Health Care and Productivity Costs | From baseline measurement to 9 months later
  Cost questionnaire developed by Health Sciences Department (Economic Evaluation) of VU University of Amsterdam

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided